CLINICAL TRIAL: NCT02073513
Title: Effects of Kinesiotaping the Hand of Children With Cerebral Palsy
Brief Title: Kinesiotaping the Hand in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, Research Assistant, MsC, PT, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUT 09/24-47
Record Dates: First submitted 2013-12-12; First posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-02

CONDITIONS: Spasticity
Keywords: Spasticity, Hand Function, Cerebral Palsy, Kinesiotape
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy | interventions — Athletic Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- kinesiotape plus thenar pressure (PPTG) (Experimental): In the kinesiotape plus thenar pressure (PPTG). Kinesiotape was applied which controled the cortical thumb sign. In addition a piece of plastazote aiming to give thenar pressure was also applied.
  The amount of pressure was regulated so that the child felt the pressure without being irritated and without restriction in grasping functions.
  Interventions: Device: Kinesiotape plus thenar pressure (PPTG)
- Taping Group (TG) (Experimental): In the taping group (TG) kinesiotape was applied to control the cortical thumb sign.
  Interventions: Device: Taping Group (TG)
- Control Group (CG) (No Intervention): No application.

INTERVENTIONS:
Device: Kinesiotape plus thenar pressure (PPTG) — In the kinesiotape plus thenar pressure (PPTG). Kinesiotape was applied to control the cortical thumb sign. In addition a piece of plastazote aiming to give thenar pressure was also applied.
  The amount of pressure was regulated so that the child felt the pressure without being irritated and without restriction in grasping functions.
  Arms: kinesiotape plus thenar pressure (PPTG)
Device: Taping Group (TG) — In the taping group (TG) kinesiotape was applied to control the cortical thumb sign.
  Arms: Taping Group (TG)

SUMMARY:
BACKROUNDS: Thumb in palm deformity restricts hand function by prevent somatosensory input in the children with cerebral palsy who have spasticity in their hands.

OBJECTİVES: To investigate the effects of thenar palmar kinesiotape application with and without pressure on hand function in children with cerebral palsy. METHOD: 45 children were randomly allocated to one of the thenar taping groups either with or without pressure or to the control group. Nine hole peg test and nine parts puzzle test were used to measure hand function. The two study groups were evaluated initially, with taping 20 minutes later and 20 minutes after taping was removed.

DETAILED DESCRIPTION:
BACKROUNDS: Thumb in palm deformity restricts hand function by prevent somatosensory input in the children with cerebral palsy who have spasticity in their hands.

OBJECTİVES: To investigate the effects of thenar palmar kinesiotape application with and without pressure on upper extremity function in children with cerebral palsy. METHOD: 45 children were randomly allocated to one of the thenar taping groups either with or without pressure or to the control group. Nine hole peg test and nine parts puzzle test were used to measure upper extremity function. The two study groups were evaluated initially, with taping 20 minutes later and 20 minutes after taping was removed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cerebral Palsy
* Stable clinical status
* Hand and/ or wrist spasticity
* No passive movement limitation
* Receiving regular neurodevelopmental rehabilitation
* Sufficient cognitive level

Exclusion criteria:

* Surgery of the upper extremity
* Orthotic treatment
* Sensory deficit

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Nine hole peg test | at baseline (before application), at 20 minutes after application, at 20 minutes after application removed

SECONDARY OUTCOMES:
nine parts puzzle test | at baseline (before application), at 20 minutes after application, at 20 minutes after application removed

CONTACTS AND LOCATIONS:
Overall Officials: Fatma UYGUR, Prof. PhD., Study Director — Hacettepe University Ethical Committee
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Ankara, Turkey (Türkiye)